CLINICAL TRIAL: NCT01135550
Title: A RANDOMIZED CONTROLLED MULTICENTER NON-INFERIORITY TRIAL OF TWICE DAILY LOW DOSE DEXAMETHASONE VERSUS USUAL DOSE DEXAMETHASONE FOR SYMPTOM CONTROL IN CHILDREN WITH A BRAIN TUMOUR UNDERGOING CRANIAL OR CRANIOSPINAL RADIATION
Brief Title: Low Dose Versus Usual Dose Dexamethasone for Symptom Control in Children Undergoing Cranial or Craniospinal Radiation
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: premature closure due to lack of accrual
Sponsor: The Hospital for Sick Children (Other)
Collaborators: C17 Council (Other)
Responsible Party: Principal Investigator, Ute Bartels, Staff Physician, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 1000014713
Record Dates: First submitted 2010-06-01; First posted 2010-06-02 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Vomiting; Headache
Keywords: Pediatrics; Vomiting; Headache; Radiation Therapy
MeSH Terms: conditions — Vomiting; Headache | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Arm (Active Comparator): Subjects scheduled to undergo radiation therapy are enrolled before the therapy is started. Once radiation therapy begins they will complete a daily diary about any headaches or nausea/vomiting they experience.
  If they experience increased headache or vomiting they will be randomized to receive either a high or a low dose of dexamethasone, to control these symptoms.
  Interventions: Drug: High dose dexamethasone
- Control Arm (Active Comparator): Subjects scheduled to undergo radiation therapy are enrolled before the therapy is started. Once radiation therapy begins they will complete a daily diary about any headaches or nausea/vomiting they experience.
  If they experience increased headache or vomiting they will be randomized to receive either a high or a low dose of dexamethasone, to control these symptoms.
  Interventions: Drug: Low dose dexamethasone

INTERVENTIONS:
Drug: High dose dexamethasone — Subject will receive 5 mg/m2 po divided in two doses. Dexamethasone 4mg/mL solution will be compounded into a 1mg/mL dosage form.
  If symptoms are well controlled over 2 weeks time, tapering of dexamethasone can be considered. It will be at the treating physician's discretion to decide the start of the tapering of dexamethasone. The weaning schedule will be the same in both intervention arms: halving the dose once weekly (week 1, week 2) while continuing to give two doses/day, one half morning dose at week 3 and every second day at week 4.
  Arms: Standard Arm
Drug: Low dose dexamethasone — Subject will receive 1 mg/m2 po divided in two doses. Dexamethasone 4mg/mL solution will be compounded into a 1mg/mL dosage form.
  If symptoms are well controlled over 2 weeks time, tapering of dexamethasone can be considered. It will be at the treating physician's discretion to decide the start of the tapering of dexamethasone. The weaning schedule will be the same in both intervention arms: halving the dose once weekly (week 1, week 2) while continuing to give two doses/day, one half morning dose at week 3 and every second day at week 4.
  Arms: Control Arm

SUMMARY:
The purpose of this study is to evaluate the effectiveness of low dose dexamethasone versus high dose dexamethasone in the treatment of radiation induced vomiting.

DETAILED DESCRIPTION:
Dexamethasone is an effective medication to ameliorate radiation induced headache and vomiting. In our Toronto experience dexamethasone in low doses (1 mg/m2/day) is sufficient in treating these symptoms. However this experience is not shared from many neuro-oncology centers of excellence that more commonly use 5 mg/m2/day according to the results of the trans-Canadian survey. A prospective multicenter trial evaluating the effectiveness of dexamethasone in different dose regimens in symptomatic children while undergoing CNS radiation will elucidate the appropriate dose.

ELIGIBILITY:
Inclusion Criteria for Enrolment:

* Children between 2-18 years of age.
* Children who underwent resection of a brain tumour with ≤ 1.5 cm2 residual tumour after surgical resection.
* Children regardless of extent of leptomeningeal or spinal metastasis (M1-3) are eligible.
* Children who undergo focal or whole brain (± spinal) radiation as part of their brain tumour treatment.
* Children treated at one of the 16 tertiary care centers in Canada (CPBTC).
* Patients on any anticonvulsive treatment are eligible.
* Patients on concomitant chemotherapy while undergoing radiation are eligible.
* Patients must be ≥ 24 hours steroid-free prior to starting radiation.
* Parents/legal guardians have to have signed and dated an informed consent to allow study enrolment of their child. (As per institutional guidelines, patients over a certain age may have signed their own informed consent form.)
* Patients > 8 years of age should assent to study participation.
* Patients less than 10 years of age should have a Lansky Score of >/= 50.
* Patients 10 years of age or older should have a Karnofsky Score of >/= 50. If ECOG performance scale is used, patient should have a score of 0, 1 or 2.

Exclusion Criteria for Enrolment:

* Children with residual brain tumour lesion > 1.5 cm2 after surgical resection.
* Children on steroids (dexamethasone) that will not be stopped ≥ 24 hours prior to start of radiation therapy.

Inclusion Criteria for Randomization to a Dexamethasone treatment group:

* Patients must have been enrolled on the Dexamethasone study prior to the start of radiation therapy.
* Children who develop either symptoms of vomiting (defined as either retching or vomiting ≥ once per day) or headache (≥ 2 points increase in severity of the most intense headache/day) while undergoing irradiation.
* Patients who are currently undergoing focal or whole brain (± spinal) radiation.

Exclusion Criteria for Randomization to a Dexamethasone treatment group:

* Patients who were not enrolled on Dexamethasone study prior to start of radiation therapy.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2010-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Effectiveness of dexamethasone on vomiting | 24-48 hours after first dose of dexamethasone
  The primary outcome will be the evaluation of effectiveness of dexamethasone on vomiting after 24-48 hours (after 2-4 doses of treatment). Vomiting is defined as either retching or vomiting and will be counted in events. The frequency of emetic episodes/day will be documented in the daily diary. The effectiveness of dexamethasone will be counted in number of episodes and evaluated on day 2 (48 hours after first dose).

SECONDARY OUTCOMES:
Headaches | 0-48 hours after first dose of dexamethasone
  Parent/patients are asked to document the worst headache of the day prior to bedtime daily on a visual analogue scale using the 6-face "happy face" scale ranging from 0 (no headache) to 5 (extreme headache).
Adverse events and side effects | Duration of participation in study
  These will be described with numbers, type and frequencies for the duration of the subjects participation in the study.
Quality of life | Baseline and at end of participation in study
  Parent/patient will complete a quality of life assessment within 14 days prior to starting radiation (including first day of radiation) and within 14 days post completion of radiation (including last day of radiation).

CONTACTS AND LOCATIONS:
Overall Officials: Ute Bartels, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (5):
- Canada (5):
  - Alberta Children's Hospital, Calgary, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - McMaster University Hospital, Hamilton, Ontario
  - Children's Hospital of Western Ontario, London, Ontario
  - The Hospital for Sick Children, Toronto, Ontario